CLINICAL TRIAL: NCT06003582
Title: Partnership for Change - Co-production and Feasibility Randomised Controlled Trial of an Intervention to Improve the Mental Health of Children With a Social Worker
Brief Title: Co-production and Feasibility RCT of Intervention to Improve the Mental Health of Children With a Social Worker
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: National Society for the Prevention of Cruelty to Children (Other); Glasgow City Council (Unknown); London Borough of Bromley (Unknown); University of Nottingham (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Helen Minnis, Professor Helen Minnis, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 316250
Record Dates: First submitted 2023-05-11; First posted 2023-08-22 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Parent-Child Relations; Child Mental Disorder; Child Maltreatment
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Infant mental health service
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant Parent Support (Experimental): Families engage with the new therapeutic intervention, Infant Parent Support.
  Interventions: Other: Infant Parent Support
- Services As Usual (No Intervention): Families randomised to Services As Usual, engage with already existing services.

INTERVENTIONS:
Other: Infant Parent Support — Therapeutic Intervention
  Arms: Infant Parent Support

SUMMARY:
Feasibility RCT to ask: Can the investigators coproduce, with parent collaborators, a new service, Infant Parent Support (IPS), to improve the mental health of children with a social worker? Can the investigators test the feasibility of an RCT of IPS compared with services as usual?

DETAILED DESCRIPTION:
Questions addressed: Can the investigators coproduce, with parent collaborators, a new service, Infant Parent Support (IPS), to improve the mental health of children with a social worker? Can the investigators test the feasibility of an RCT of IPS compared with services as usual?

Considered for entry: Parents of children aged 0-5 who have mental health concerns, social workers, and a multi-agency support plan.

Inclusion criteria: Any family in the Glasgow or Bromley trial sites with a child aged 0-5 years with mental health concerns, a social worker, and a multi-agency support plan.

Exclusion criteria: At the outset of the Trial there were no exclusion criteria.

Over the course of Phase 1, the following exclusion criteria have emerged:

* If the child has a Child Protection Plan or is on the Child Protection Register
* If the family are in the process of 'stepping down' from a CPP or CPR
* If the child is currently engaged in therapeutic work.

Intervention: Infant Parent Support (a multidisciplinary infant mental health team aiming to improve the mental health of children aged 0-5 with a social worker).

Primary Outcomes Phase 1: Coproduction, with parents of children who have a social worker, of the IPS intervention.

Phase 2: Recruitment and retention (at 3 and 6 months) to a feasibility RCT.

Secondary Outcomes

Phase 1: preliminary mapping of service context.

Phase 2:

* Improvement in the organisation, access, and quality of services, for children with a social worker and mental health issues.
* Examination of putative primary and secondary outcomes for a future definitive RCT of IPS (see below)
* Development of a parent-supported outcome measure and a parent-supported experience measure for use in a future definitive RCT
* Exploration of whether it is possible to expand into new sites to conduct a successful Phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Any family in the Glasgow or Bromley trial sites with a child aged 0-5 years with mental health concerns, a social worker, and a multi-agency support plan.

Exclusion Criteria:

At the outset of the Trial there were no exclusion criteria. Over the course of Phase 1, the following exclusion criteria have emerged:

* If the child has a Child Protection Plan or is on the Child Protection Register
* If the family are in the process of 'stepping down' from a CPP or CPR
* If the child is currently engaged in therapeutic work.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates to a feasibility RCT | 6 months
  The recruitment of 30 families to the Trial and the 15 families randomised to the new therapeutic intervention will be measured by recruitment rates.
Retention rates to a feasibility RCT | 1 year
  The proportion of the 15 families randomised to the new intervention who continue through the Trial will be measured by retention rates.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Minnis, PhD, Principal Investigator — University of Glasgow
Locations (1):
- London Borough of Bromley, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pownall J, Crawford K, Dalgarno L, Fisher J, Graham S, Turner F, Minnis H, Boyd K, Seyahian A, McConnachie A, Cosgrave N, Forde M, Atkinson C, McCullough J, Sayal K, Ougrin D. Infant Parent Support (IPS): a multidisciplinary intervention to improve the mental health of children with a social worker - a study protocol for a feasibility randomised controlled trial with embedded process evaluation. Pilot Feasibility Stud. 2025 Jun 5;11(1):78. doi: 10.1186/s40814-025-01616-6. PMID 40474316